CLINICAL TRIAL: NCT03041545
Title: Tracking Physical Activity Throughout Chemotherapy for Breast Cancer
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Sheri Hartman, Assistant Professor, University of California, San Diego
Other Study IDs: 150860; 5U54CA155435-05 (NIH)
Record Dates: First submitted 2017-01-30; First posted 2017-02-02 (Estimated); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Breast Cancer; Physical Activity
MeSH Terms: conditions — Breast Neoplasms; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fitbit: All participants will be asked to wear the Fitbit as much as possible and to sync it at least once a week, from one week prior to start of chemotherapy treatment to six months after ending chemotherapy.
  Interventions: Device: Fitbit

INTERVENTIONS:
Device: Fitbit — Women enrolled in the study will be asked to wear a Fitbit from one week prior to chemotherapy until six months post-chemotherapy. The Fitbit is a watch-sized, wrist worn, physical activity tracker. A button, when pressed, displays the wearer's accumulated daily steps, mileage, and steps climbed.

SUMMARY:
Physical activity during chemotherapy has been shown to increase patient health and wellbeing as well as improve outcomes in breast cancer patients. The primary aim of this project is to determine the feasibility of incorporating wearable sensors into clinical care by having breast cancer patients, undergoing chemotherapy, wear a commercially available monitor (Fitbit) that tracks physical activity, sleep, and heart rate monitor.

DETAILED DESCRIPTION:
Although there are many benefits of engaging in physical activity during cancer treatments, activity levels typically decline throughout treatment. Existing research has primarily relied on self-reported activity levels and only captured periodic snap shots or retrospective reports of activity levels, which are subject to recall bias. Exactly how activity levels change throughout chemotherapy is not known. This study will provide minute-by-minute level objective physical activity data across the entirety of the patient's chemotherapy treatments. This in depth data will provide a new perspective on the patterns of activity levels and help to identify if there are critical times in which to intervene to prevent declines in physical activity.

The investigators will assess the feasibility of the pre-treatment recruitment by documenting recruitment rates and participant acceptance of wearing the accelerometer.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Diagnosed with breast cancer
* Scheduled to receive chemotherapy, but has not yet started chemotherapy
* Receiving chemotherapy at a University of California, San Diego clinic
* Willingness to wear the Fitbit throughout the course of chemotherapy
* Access to a computer or Bluetooth enabled phone to sync Fitbit data
* Able to read and communicate in English

Exclusion Criteria:

• Serious physical limitation that greatly limits mobility

Ages: 21 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is all women approached to attempt recruitment. Women will be recruited through the Medical Oncology Clinics at UCSD Moroes Cancer Center.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2018-02-08 (Actual); Study Completion 2018-02-08 (Actual)

PRIMARY OUTCOMES:
Recruitment | 06/01/2015-06/01/2018
  Enrolling >20% of eligible patients

SECONDARY OUTCOMES:
Retention | From date enrolled into the study until 1 week after the date of the last infusion center visit for chemotherapy, which is typically up to 6 months.
  >80% of participants wore the Fitbit for >80% of the days during chemotherapy treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sheri J Hartman, PhD, Principal Investigator — Assistant Professor
Locations (1):
- University of California, San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No